CLINICAL TRIAL: NCT05501028
Title: Using Natural Language Processing of Novel Biopsychosocial Disease Constructs to Aid in the Evaluation and Diagnosis of Functional Gastrointestinal Disorders
Brief Title: NLP to Aid in the Evaluation and Diagnosis of FGIDs
Status: Enrolling by invitation | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Kyle Staller, MD, MPH, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2018P001542
Record Dates: First submitted 2022-03-01; First posted 2022-08-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients scheduled for consult with gastroenterologist
- Patients scheduled for diagnostic endoscopy

SUMMARY:
The study has two arms, where the same natural language processing (NLP) and probabilistic graphical modeling technology will be utilized on patients' report of symptoms in both arms. The clinical arm is focused on patients presenting for consultation with a gastroenterologist. The endoscopy arm is focused generally on patients presenting for a diagnostic endoscopy, with the goal of capturing Functional Gastrointestinal Disorder (FGID) patients prior to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for consult in the Motility Clinic in the MGH Gastroenterology Unit or for diagnostic endoscopy in the MGH Gastroenterology Unit
* Patient must agree to have their interactions audio-recorded
* Informed consent form signed by the subjects

Exclusion Criteria:

* Non-native English speaker
* Patients unable to communicate their own symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients who are scheduled for a consult in the MGH Gastroenterology Unit
  Group 2: Patients who are scheduled for a diagnostic endoscopy in the MGH Gastroenterology Unit
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Latent themes present in patient descriptions of FGIDs symptoms | 08/09/2018-08/09/2023
  Latent themes present in patient descriptions of FGIDs symptoms as generated by machine learning as well as quantitative comparisons to traditional metrics of patient descriptions including Rome IV criteria and patient descriptions of severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided